CLINICAL TRIAL: NCT00717314
Title: A Randomized, Open Label Study Comparing the Effect of CellCept Combined With 2 Regimens of Reduced Calcineurin Inhibitors on Kidney Function in Liver Transplant Patients
Brief Title: A Study of CellCept (Mycophenolate Mofetil) Combined With Calcineurin Inhibitors in Liver Transplant Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21241
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Mycophenolic Acid; cni protein, Drosophila

ARMS (2):
- MMF, 50% CNI Reduction (Experimental): Participants received mycophenolate mofetil (MMF), 1.5 to 2.0 grams (g) daily, orally (PO), twice per day (BID) from baseline (BL) to Week 52. Participants also received a 50 percent (%) reduced dose of calcineurin inhibitor (CNI) from BL to Week 52.
  Interventions: Drug: Mycophenolate mofetil; Drug: CNI (50%)
- MMF, ≥75% CNI Reduction (Experimental): Participants received MMF, 1.5 to 2.0 g daily, PO, BID from BL to Week 52. Participants also received a 75% reduced dose of CNI from BL to Week 52.
  Interventions: Drug: Mycophenolate mofetil; Drug: CNI (≥75%)

INTERVENTIONS:
Drug: Mycophenolate mofetil — 1.5 to 2.0 g daily PO BID
  Other Names: CellCept
Drug: CNI (50%) — 50% reduction from BL
  Arms: MMF, 50% CNI Reduction
Drug: CNI (≥75%) — ≥75% reduction from BL
  Arms: MMF, ≥75% CNI Reduction

SUMMARY:
This 2 arm study will compare the efficacy and safety of switching to CellCept combined with different regimens of reduced calcineurin inhibitors (CNI) in patients with liver transplants. Patients currently receiving CNI treatment will be randomized into one of 2 groups to receive either 1) CellCept 2.0g/day po bid + 50% reduction of CNI from baseline or 2) CellCept 2.0g/day po bid + >=75% reduction of CNI from baseline. The anticipated time on study treatment is 1 year, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* single organ recipients of liver allograft;
* CNI-based immunosuppressive regimen prior to study entry and regimen adjustment;
* >=6 months post-transplant, with renal dysfunction (serum creatinine 140-300micromol/L at entry);
* negative pregnancy test for women of childbearing potential; contraception must be taken before beginning study drug therapy and until 6 weeks after last dose of study medication.

Exclusion Criteria:

* treatment with CellCept or any other product which delivers mycophenolic acid within the 3 months prior to the recent switch to CellCept relevant for enrollment;
* known contraindications to CNI, corticosteroids or CellCept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- China (9):
  - Beijing
  - Changsha
  - Chengdu
  - Chongqing
  - Guangzhou
  - Jiangsu
  - Shanghai
  - Tianjin
  - Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil (MMF), 50% Calcineurin Inhibitor (CNI): Participants received MMF capsules, 1.5 to 2.0 grams (g), orally (PO), twice daily (BID) up to Week 52. Participants also received a CNI (at discretion of investigator) at a reduced dosage of up to 50 percent (%) through Week 52. The dosage of CNI was reduced to 25% of the dose at entry within the first week, and to 50% of the dose at entry within the first 2 weeks. This 50% reduced CNI dose was to be continued through Week 52. Corticosteroids were administered per documented center practice throughout the study with a goal of reducing steroid dose to 0 by 13 weeks post-transplant.
- MMF, 75% CNI: Participants received MMF capsules, 1.5 to 2.0 g, PO, BID up to Week 52. Participants also received a CNI (at discretion of investigator) at a reduced dosage of up to at least 75% through Week 52. The dosage of CNI was reduced to 50% of the dose at entry within the first 2 weeks, and to at least 75% of the dose at entry within the following 2 weeks. This 75% reduced CNI dose was to be continued through Week 52. Corticosteroids were administered per documented center practice throughout the study with a goal of reducing steroid dose to 0 by 13 weeks post-transplant.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil (MMF), 50% Calcineurin Inhibitor (CNI) | MMF, 75% CNI
Started | 43 | 44
Completed | 37 | 34
Not Completed | 6 | 10
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 5
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: Per-Protocol (PP) population: all participants who received at least 1 dose of the treatment-group specific medication who did not dropout from the study prematurely.
Groups:
- MMF, 50% CNI: Participants received MMF capsules, 1.5 to 2.0 g, PO, BID up to Week 52. Participants also received a CNI (at discretion of investigator) at a reduced dosage of up to 50% through Week 52. The dosage of CNI was reduced to 25% of the dose at entry within the first week, and to 50% of the dose at entry within the first 2 weeks. This 50% reduced CNI dose was to be continued through Week 52. Corticosteroids were administered per documented center practice throughout the study with a goal of reducing steroid dose to 0 by 13 weeks post-transplant.
- Total: Total of all reporting groups
Arm/Group | MMF, 50% CNI | MMF, 75% CNI | Total
Number analyzed (Participants) | 37 | 34 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (8.7) | 52.4 (11.1) | 52.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — PP population included all participants completing study treatment, n= 37 and 34 participants in the MMF, 50% CNI Reduction and MMF, ≥75% CNI Reduction groups, respectively.
  Participants
    Female | 4 | 4 | 8
    Male | 33 | 30 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Decrease in Glomerular Filtration Rate (GFR) of Greater Than 20%
Description: The percentage of participants with a greater than 20% decrease of GFR during the 1-year period following regimen adjustment. Cockcroft and Gault formula was used for calculated creatinine clearance.
Time Frame: Week 52
Population: PP population
Measure: Number; unit: percentage of participants
Arm/Group | MMF, 50% CNI | MMF, 75% CNI
Number analyzed (Participants) | 37 | 34
percentage of participants | 5.4 | 0.0
Statistical Analysis 1: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Test type: Superiority or Other; p = 0.494, ANOVA

2. Secondary Outcome: Percentage of Participants With Graft Loss or Death at Week 52
Description: Graft loss was defined for this protocol as re-transplantion or death.
Time Frame: Week 52
Population: PP population
Measure: Number; unit: percentage of participants
Arm/Group | MMF, 50% CNI | MMF, 75% CNI
Number analyzed (Participants) | 37 | 34
percentage of participants
  Graft loss | 0.0 | 0.0
  Death | 0.0 | 0.0

3. Secondary Outcome: Percentage of Participants With Biopsy-Proven Acute Rejection (BPAR) at Week 52
Description: BPAR was graded according to Banff criteria.
Time Frame: Week 52
Population: PP population
Measure: Number; unit: percentage of participants
Arm/Group | MMF, 50% CNI | MMF, 75% CNI
Number analyzed (Participants) | 37 | 34
percentage of participants | 0.0 | 5.9

4. Secondary Outcome: Changes From Baseline in Creatinine Clearance (Milliliters Per Minute [mL/Min])
Description: Creatinine clearance calculated using the Cockcroft and Gault formula: For adult males, creatinine clearance in mL/min equaled (=) [(140 minus (-) age in years) multiplied by (*) (weight in kilograms (kg)] divided by [72 * serum creatinine in milligrams per deciliter (mg/dL)]. For adult females, creatinine clearance in mL/min = 0.85 * [(140 - age in years) * (weight in kg)] divided by (72 * serum creatinine in mg/dL).
Time Frame: Baseline and Weeks 16, 28, and 40
Population: PP population; number (n) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | MMF, 50% CNI | MMF, 75% CNI
Number analyzed (Participants) | 37 | 34
mL/min
  Baseline (n=36,31) | 1.385 (3.433) | 2.250 (4.469)
  Change at Week 16 (n=37,33) | 4.884 (6.016) | 5.629 (8.825)
  Change at Week 28 (n=34,33) | 5.333 (9.365) | 4.560 (8.325)
  Change at Week 40 (n=35,27) | 6.131 (9.148) | 4.125 (10.802)
Statistical Analysis 1: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Between group comparison at Baseline; Test type: Superiority or Other; p = 0.374, ANOVA
Statistical Analysis 2: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Change from Baseline at Week 16; Test type: Superiority or Other; p = 0.685, ANCOVA — Analysis of covariance (ANCOVA) model with calculated creatinine clearance at baseline as covariate, and study center and treatment*study center as factors
Statistical Analysis 3: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Change from Baseline at Week 28; Test type: Superiority or Other; p = 0.722, ANCOVA — ANCOVA model with calculated creatinine clearance at baseline as covariate, and study center and treatment*study center as factors
Statistical Analysis 4: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Change from Baseline at Week 40; Test type: Superiority or Other; p = 0.432, ANCOVA — [p-value comment as in outcome 4, analysis 3]

5. Secondary Outcome: Change From Baseline in Corrected Creatinine Clearance (mL/Min) at Week 52
Description: Corrected creatinine clearance was calculated using the Cockcroft and Gault formula: For adult males, creatinine clearance in mL/min = [(140 - age in years) * (weight in kg] divided by [72 * serum creatinine in mg/dL]. For adult females, creatinine clearance in mL/min = 0.85 * [(140 - age in years) * (weight in kg)] divided by (72 * serum creatinine in mg/dL).
Time Frame: Week 52
Population: PP population; number (n) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | MMF, 50% CNI | MMF, 75% CNI
Number analyzed (Participants) | 37 | 34
mL/min | 6.551 [2.850 to 10.253] | 6.442 [2.575 to 10.309]
Statistical Analysis 1: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Test type: Superiority or Other; Mean Difference (Final Values) = 0.110, 95% CI 2-sided [-5.342 to 5.561]

6. Secondary Outcome: Percentage Change in Creatinine Clearance From Baseline
Description: Creatinine clearance was calculated using the Cockcroft and Gault formula.
Time Frame: Weeks 16, 28, 40, and 52
Population: PP population
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | MMF, 50% CNI | MMF, 75% CNI
Number analyzed (Participants) | 37 | 34
percentage change from baseline
  Week 16 (n=37,33) | 10.38 (13.97) | 8.72 (13.45)
  Week 28 (n=34,33) | 11.45 (19.87) | 7.51 (12.53)
  Week 40 (n=35,27) | 12.37 (19.14) | 7.03 (17.86)
  Week 52 (n=37,34) | 10.17 (20.63) | 11.51 (16.20)
Statistical Analysis 1: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Change from Baseline at Week 16; Test type: Superiority or Other; p = 0.616, ANCOVA — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 2: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Change from Baseline at Week 28; Test type: Superiority or Other; p = 0.334, ANCOVA — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 3: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Change from Baseline at Week 40; Test type: Superiority or Other; p = 0.267, ANCOVA — [p-value comment as in outcome 4, analysis 3]
Statistical Analysis 4: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Change from Baseline at Week 52; Test type: Superiority or Other; p = 0.764, ANCOVA; ANCOVA model with calculated creatinine clearance at baseline as covariate, and study center and treatment*study center as factors

7. Secondary Outcome: Percentage of Participants Experiencing Acute Rejection, Graft Loss, Death, or a Decrease From BL in Creatinine Clearance of ≥20% at Week 52
Description: The percentage of participants who experienced at least 1 of the following: a ≥20% decrease from BL in creatinine clearance, acute rejection, graft loss, or death 1 year after randomization.
Time Frame: Week 52
Population: PP population
Measure: Number; unit: percentage of participants
Arm/Group | MMF, 50% CNI | MMF, 75% CNI
Number analyzed (Participants) | 37 | 34
percentage of participants | 8.1 | 8.8
Statistical Analysis 1: Comparison: MMF, 50% CNI vs MMF, 75% CNI; Test type: Superiority or Other; p = 1.000, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported at throughout the 52 weeks of the study. Serious AEs (SAEs) were to be reported up to 30 days after stopping the treatment or during the follow-up period; related SAEs should have continued to be reported.
Description: All participants who received at least 1 dose of study treatment were included in the safety analysis population.
Arm/Group | MMF, 50% CNI | MMF, 75% CNI
Serious Adverse Events (participants affected / at risk) | 1/43 | 3/40
Other Adverse Events (participants affected / at risk) | 15/43 | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF, 50% CNI (N=43) | MMF, 75% CNI (N=40)
Lung Infection (Infections and infestations) | 1 | 0
Acute rejection (Immune system disorders) | 0 | 1
Biliiary tract infection (Infections and infestations) | 0 | 1
Recurrent hepatitis B virus (Infections and infestations) | 0 | 1
Hepatic cancer bladder metastasis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF, 50% CNI (N=43) | MMF, 75% CNI (N=40)
Alanine aminotransferase increased (Investigations) | 1 | 4
White blood cell count decreased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3
Blood creatinine increased (Investigations) | 2 | 2
Blood urine present (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 0 | 1
Gamma-glutamytransferase increased (Investigations) | 0 | 1
Glucose urine present (Investigations) | 0 | 1
Neutrophil cound decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Urine leukocyte esterase positive (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Perihepatic discomfort (Hepatobiliary disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal injury (Renal and urinary disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.